CLINICAL TRIAL: NCT00913757
Title: A Study of Molecular and Genetic Factors for Liver Cancer in the Greater Baltimore Area
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909149; 09-C-N149; NCT00980564 (obsolete NCT alias)
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma, Hepatocellular; Liver Cirrhosis, Alcoholic; Hepatitis, Alcoholic; Hepatitis, Chronic; Hepatitis, Viral, Human
Keywords: Hepatocellular Carcinoma; Liver Cancer; Chronic Liver Disease; Genome Wide Association Study; Gene Expression Profiling
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis, Alcoholic; Hepatitis, Alcoholic; Hepatitis, Chronic; Hepatitis, Viral, Human; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples, mouth wash and urine.

GROUPS / COHORTS (3):
- Group 1: 400 patients with primary HCC (Hepatocellular carcinoma)
- Group 2: 800 patients with chronic liver disease (high risk non-cancer cases)
- Group 3: 800 population-based controls, identified through a OMV database that will match cases by age, gender, race, and county of residency

SUMMARY:
Background:

* Liver cancer is the third most deadly and fifth most common cancer worldwide. Hepatocellular carcinoma (HCC) is the most frequent primary liver cancer, and it has grown more prevalent in the United States.
* More information is needed about the causes and effects of liver cancer, and further research into individuals who are at high risk for developing liver cancer is needed for early diagnosis and prevention.

Objectives:

* To identify genetic factors that may help to explain the aggressiveness of liver cancer.
* To determine if HCC biomarkers exist in blood, urine, and tissue samples.

Eligibility:

* Patients between the ages of 18 and 90 who have been diagnosed with HCC or have a high risk for developing HCC because of fatty liver disease (alcohol-related or non-alcohol-related) or chronic hepatitis B or C.
* Participants will reside in Baltimore City and the surrounding areas.

Design:

* Participants will complete a questionnaire and provide blood and urine samples for testing:
* The questionnaire will include questions about individual and family medical history, tobacco use, and exposure to known factors for liver cancer.
* Blood and urine samples will be collected from all participants after the questionnaire.
* Tumor tissue and healthy tissue will be collected from selected participants if they undergo surgery for their cancer or disease.
* No specific treatment will be offered as part of this protocol, but participants have the option to be treated under different protocols.

DETAILED DESCRIPTION:
BACKGROUND:

Liver cancer is the third most deadly and fifth most common cancer worldwide. Hepatocellular carcinoma (HCC) is the most frequent primary cancer of the liver with rising incidence in the United States. HCC patients have a dismal outcome and are an underserved cancer population. We are proposing a liver cancer case-control and case-case study to be conducted in Baltimore, Maryland.

OBJECTIVES:

Our research is aimed to identify genetic and genomic changes that might explain the aggressive nature of liver cancer. We will test the primary hypothesis that HCC biomarkers exist in blood products (or mouth wash), urine and/or tissues that can be used for early diagnosis and prevention. A unique study factor is the use of urine samples for biomarker identification. A secondary goal will be to examine whether certain genetic and genomic factors modify liver cancer susceptibility using candidate and genome wide association study approaches. Although other studies have investigated genetic susceptibility, large scale studies have not been conducted for liver cancer. Our study will also be valuable due to access to frozen tumor specimens from pre-therapy resection, whose collection is required for gene expression analysis. If certain genes are related to HCC risk and progression, this tissue resource will be used to further validate our findings with laboratory investigations. The proposed study is designed to be exploratory and hypothesis generating.

ELIGIBILITY:

The participants will reside in Baltimore City and surrounding areas. Cases will have pathologically confirmed liver cancer or risk factors for HCC development. Risk factors include chronic liver disease due to hepatitis B and/or C viral infection, nonalcoholic steatohepatitis or alcoholic cirrhosis. The study will be supported by an epidemiological infrastructure developed by our University of Maryland School of Medicine resource contractor for ongoing lung and prostate cancer case-control studies. The enrollment of controls will begin concurrently with case accrual, and will continue for 5 years. Population-based controls will be recruited using a triple eligibility criterion, such that controls eligible for the lung/prostate study will be asked to complete a supplemental questionnaire for the liver study.

DESIGN:

The study will include 400 primary HCC cases, 800 patients with chronic liver disease (high risk non-cancer cases) and a sample of 800 population-based controls. The HCC and high risk non-cancer cases will be recruited at two Baltimore hospitals, the Veterans Affairs Medical Center, and the University of Maryland School of Medicine over a period of 13-15 years. Controls will be identified through a Department of Motor Vehicle database and match cases by age, gender, race and county of residency. The study will involve administration of a questionnaire and collection of blood (or mouth wash) from all study subjects. Fresh-frozen tumor and tumor surrounding non-cancerous specimens will be obtained from approximately 20 percent of the cancer patients. The cases will receive one questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:

SELECTION OF CASE SUBJECTS (HCC AND HIGH RISK NON-CANCER CASES)

We will recruit incident cases of pathologically confirmed primary liver cancer or risk factors for liver cancer (patients with chronic liver disease due to hepatitis B and/or C viral infection, nonalcoholic steatohepatitis or alcoholic cirrhosis) at all stages of the disease that are age greater than or equal to 18 years or less than or equal to 90 years. Treatment can be surgery or therapy. The following check list will be used to verify eligibility of a case subject.

ELIGIBILITY CRITERIA- HCC CANCER CASES

1. Diagnosed with primary liver cancer (HCC) within the last two years
2. Physician diagnosis based on AFP and ultrasound/imaging or Pathological diagnosis of primary liver cancer made at the local hospital pathology department
3. Resides in Maryland or surrounding states
4. Has a residential working phone within his/her home (*The reason for a participant having a residential working phone is that the matching population controls are selected through the Department of Motor Vehicles records and must have a residential telephone number to be selected as part of the random sample.)
5. Age is greater than or equal to 18 years and less than or equal to 90 years
6. A non-objection statement by the physician from the hospital where the patient was identified, or listed as the treating physician by the tumor registry or surgical pathology report, to contact the patient is obtained
7. Is not currently residing in an institution, such as a prison, nursing home, or shelter
8. Is not a severely ill patient in the intensive care unit
9. Is able to give informed consent
10. Is physically and mentally capable of performing the interview
11. Must understand English well enough to be interviewed
12. Has never been interviewed as a control for this study
13. Subject provides informed consent and signs form.

ELIGIBITY CRITERIA HIGH RISK NON-CANCER CASES

1. Has been diagnosed with chronic Hepatitis B or C, NASH or alcoholic liver disease with chronicity present at least for a 6 month period
2. Resides in Maryland or surrounding states
3. Has a residential working phone within his/her home
4. Age greater than or equal to 18 years and less than or equal to 90 years
5. A non-objection statement by the physician from the hospital where the patient was identified or is being treated or by the surgical pathology report, to contact the patient is obtained
6. Is not currently residing in an institution, such as a prison, nursing home, or shelter
7. Is not a severely ill patient in the intensive care unit
8. Is able to give informed consent
9. Is physically and mentally capable of performing the interview
10. Must understand English well enough to be interviewed
11. Has never been interviewed as a control for this study
12. Subject provides informed consent and signs form.

SELECTION OF POPULATION-BASED CONTROLS

Population-based controls will be identified through the Motor Vehicle Administration (MVA), and matched on age (year of birth), race, gender and geography to cases. We sample controls in proportion to the population size of their county of residence. Recruitment of controls will start concurrently with case accrual, using the age, race and gender frequency distribution of cancer patients in previous years. The sampling frame is continually updated as we accrue information on the case distribution of age, race and gender. We will exclude controls that do not have a listed home phone number. The following check list will be used to verify eligibility of a control subject.

ELIGIBILITY CRITERIA - POPULATION-BASED CONTROLS

1. Resides in Baltimore City, Anne Arundel, Baltimore, Caroline, Carroll, Cecil, Dorchester, Harford, Howard, Kent, Queen Anne s, Somerset, Talbot, Wicomica and Worchester County.
2. Has a residential working phone within his/her home
3. Age greater than or equal to 18 years and less than or equal 90 years
4. Have never had radiation therapy or chemotherapy
5. Is not currently residing in an institution, such as a prison, nursing home, or shelter
6. Is physically and mentally capable of performing the interview
7. Must understand English well enough to be interviewed
8. Has never been interviewed as a control for the study
9. Subject provides informed consent and signs form.

EXCLUSION CRITERIA:

Exclusion Criteria-HCC CANCER CASES

1. Liver cancer patients who are older than 90 years are excluded because of co-morbidity considerations and the difficulty of matching those cases with population-based controls.
2. Children and institutionalized patients are excluded from the proposed study. Very few HCC patients at the 3 participating hospitals are younger than 18 years of age and HCC incidence mainly occurs in adults.

Exclusion Criteria-HCC HIGH-RISK NON-CANCER CASES

1. High Risk Non-Cancer patients who are older than 90 years are excluded because of co-morbidity considerations and the difficulty of matching those cases with population-based controls.
2. Children and institutionalized patients are excluded from the proposed study. Very few HCC patients at the 3 participating hospitals are younger than 18 years of age and HCC incidence mainly occurs in adults. High-Risk Non-Cancer cases who are younger than 18 years are excluded due to the need of matching with HCC cases and population controls.

Exclusion Criteria-POPULATION BASED CONTROLS

1. Population based controls who are older than 90 years are excluded because of co-morbidity considerations and the difficulty of matching with HCC cases and high risk non-cancer cases.
2. Population controls who are younger than 18 years or are institutionalized are excluded due to the need of matching with HCC cases and high-risk non-cancer cases.
3. Population controls with prior cancer with the exception of non-melanomic skin cancer (squamous or basal cell).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 400 primary HCC cases, 800 patients with chronic liver disease (high risk non-cancer cases) and a sample of 800 population-based controls. The HCC and high risk non-cancer cases will be recruited at two Baltimore hospitals, the Veterans Affairs Medical Center and the University of Maryland School of Medicine over a period of 13 - 15 years. Controls will be identified through a Department of Motor Vehicle database and match cases by age, gender, race and county of residency.
Sampling Method: Non-Probability Sample
Enrollment: 1871 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Large-scale molecular profiling study to identify HCC biomarkers for early diagnosis and prevention. | ongoing
  Identification of HCC biomarkers for early diagnosis and prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center, Baltimore, Maryland